CLINICAL TRIAL: NCT01281761
Title: Phase II Simvastatin + Cetuximab/Irinotecan in K-ras Mutant Colorectal Cancer Patients Who Have Failed Irinotecan and Oxaliplatin-based Chemotherapy
Brief Title: Simvastatin + Cetuximab/Irinotecan in K-ras Mutant Colorectal Cancer (CRC)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Won Ki Kang, Professor, Samsung Medical Center
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SMC IRB 2010-08-006
Record Dates: First submitted 2011-01-20; First posted 2011-01-24 (Estimated); Last update posted 2013-06-14 (Estimated); Status verified 2013-06

CONDITIONS: Metastatic Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Cetuximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- cetuximab/irinotecan/simvastatin (Experimental): D1 Cetuximab 500mg/m2 IV stepwise shortened infusion duration- [C1D1 over 120min, C2D1 over 90min,subsequent dose over 60min] D1 Irinotecan 150-180mg/m2 + Dextrose 5% 500ml IV [over 90min] D1-14 Simvastatin 80mg P.O(continuous, daily)
  * every 2weeks
  Interventions: Drug: cetuximab/irinotecan/simvastatin

INTERVENTIONS:
Drug: cetuximab/irinotecan/simvastatin — D1 Cetuximab 500mg/m2 IV stepwise shortened infusion duration- [C1D1 over 120min, C2D1 over 90min,subsequent dose over 60min] D1 Irinotecan 150-180mg/m2 + Dextrose 5% 500ml IV [over 90min] D1-14 Simvastatin 80mg P.O(continuous, daily) every 2weeks

SUMMARY:
Based on the results from preclinical study, the investigators suggest that the addition of simvastatin at a dose of cardiovascular use (40 ~ 80 mg qd daily) may overcome cetuximab resistance in KRAS mutant colorectal cancer via B-Raf protein degradation and inducing Bim and Bad. Given the result of a phase II FOLFIRI plus cardiovascular dose of simvastatin (80mg qd daily) and this study, phase II study of conventional cetuximab treatment with 40 mg simvastatin is planned in metastatic colorectal cancer patients with KRAS mutation.

DETAILED DESCRIPTION:
Simvastatin is a 3-hydroxy-3-methylglutaryl coenzyme A (HMG-CoA) reductase inhibitor leading to inhibition of post-translational modification of small G proteins. Mevalonate-derived prenyl groups, farnesyl pyrophosphate (FPP) and geranylgeranyl pyrophosphate (GGPP), facilitate essential intracellular functions of various proteins such as Ras and Rho. Owing to its effect on post-transcriptional modifications of Ras and Rho, the anti-tumor effect of statins has been suggested in various cancer cell lines. However, more recent studies utilizing cancer gene signatures have systematically screened an array of drugs for potential anti-tumor effect and have discovered statins as potential novel targeted agent against cancer. Given the cardiovascular therapeutic dose is 1 mg/kg/day which translates into serum level of 0.1 uM in patients, the investigators have previously tested and reported that low dose lovastatin ranging from nanomolar to 0.3- 1 uM statin induced cell senescence or cytostatic effect of prostate cancer cells in vitro. In addition, the investigators previously reported on well tolerability and promising anti-tumor effect of combination of simvastatin 40 mg daily and standard FOLFIRI (irinotecan, infusional 5-fluorouracil, leucovorin) in metastatic colorectal cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically-confirmed, advanced/metastatic colorectal carcinoma Failed both oxaliplatin and irinotecan based regimens for advanced/metastatic disease (last regimen has to be irinotecan-based chemotherapy; To be eligible, patients must also have received one of several qualifying, irinotecan regimens for at least 6 weeks and must have had documented progression of disease during receipt of this regimen or within six months thereafter.
2. Ras mutation (+) (checked at the central lab)
3. At least one measurable tumor mass according to RECIST 1.1
4. Expected survival for approximately 12 weeks or longer
5. Karnofsky Performance Score (KPS) ≥ 70
6. Age ≥ 18 years
7. WBC ≥ 3,500 cells/mm3 and ≤ 50,000 cells/mm3
8. ANC ≥ 1,500 cells/mm3
9. Hemoglobin ≥ 10 g/dL (transfusion allowed)
10. Platelet count ≥ 100,000 plts/mm3
11. Total bilirubin ≤ 1.5ULN
12. AST, ALT ≤ 2.5 ULN (if liver metastases(+): AST,ALT ≤5.0 x ULN)
13. Serum chemistries within normal limits (WNL) or Grade 1 (excluding alkaline phosphatase) - If patients are diabetic or have a screening random glucose > 160 mg/dL, a fasting glucose must be done and patients must be WNL or Grade 1 in order to be eligible for the study.
14. Written informed consent

Exclusion Criteria:

1. Prior simvastatin therapy within 1-year from the date of study entry
2. Severe or unstable cardiac disease, including (for example) coronary artery disease requiring increased doses of anti-anginal mediation and/or coronary angioplasty (including stent placement) within the preceding 24 months
3. Current, known CNS malignancy (history of completely resected or irradiated brain metastases by WBRT or stereotactic radiosurgery allowed)
4. Patients with CPK > 5 x ULN at baseline
5. Patients with alcohol abuse
6. Uncontrolled hypothyroidism
7. Concomitant use with clarithromycin, erythromycin, itraconazole, ketoconazole, nefazodone, telithromycin
8. Concomitant use of gemfibrozil, cyclosporine, danazol, amiodarone, verapamil

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2010-11; Primary Completion 2012-09 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
response rate | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Won Ki Kang, MD, Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea